CLINICAL TRIAL: NCT07156266
Title: Comparative Effects of Kegal and Squat Exercises on Urinary Incontinence Severity and Quality of Life
Brief Title: Comparative Effects of Kegal vs Squat Exercises on Urinary Incontinence Severity and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Dr Izza Ayub; PT, Lecturer, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUF/PB/45/1038/45
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Kegal Exercise Group) (Experimental)
  Interventions: Procedure: Kegal Exercise
- Group B (Squats Exercise Group) (Active Comparator)
  Interventions: Procedure: Squats Exercise

INTERVENTIONS:
Procedure: Kegal Exercise — Dead Bugs:Participants will begin by lying on their backs with their arms extended overhead and legs bent at a 90-degree angle. While engaging their core muscles, they will gradually lower their arms and legs toward the floor, then return to the starting position.
  Bridging Exercise: Lying on their backs with knees bent and feet flat on the ground, participants will gently raise their hips upward while activating the pelvic floor muscles, then slowly lower them back to the starting position.
  Arms: Group A (Kegal Exercise Group)
Procedure: Squats Exercise — Sumo Squats: Participants will stand with their feet placed wider than shoulder-width apart and toes pointing outward. They will then squat down, keeping their backs straight and their weight on their heels, pause briefly at the bottom, and return to a standing position.
  Narrow Squats: With their feet set shoulder-width apart and toes pointing forward or slightly outward, participants will lower their bodies into a squat position while keeping their backs straight and their weight centered in the heels. After a brief pause, they will return to a standing position.
  Arms: Group B (Squats Exercise Group)

SUMMARY:
A randomized clinical trial will be carried out to compare the effectiveness of Kegel and squat exercises in reducing urinary incontinence. The study will include 30 participants diagnosed with urinary incontinence, who will be randomly assigned to either a Kegel exercise group or a squat exercise group. Both groups will perform their respective exercises for 10 minutes, three times daily, over a period of 12 weeks. Outcomes will be assessed using the International Consultation on Incontinence Questionnaire - Female Lower Urinary Tract Symptoms Long Form (ICIQ-FLUTS LF) and the Incontinence Quality of Life (I-QOL) questionnaire

ELIGIBILITY:
Inclusion Criteria Women aged between 30 and 60 years with a confirmed diagnosis of urinary incontinence (UI) by a qualified healthcare professional.

Women who are physically able to perform the required exercises and are willing to provide informed consent to participate in the study.

Exclusion Criteria

Pregnant women or those planning to become pregnant during the study period. Individuals who have undergone surgery within the past six months that may affect pelvic floor strength or urinary incontinence symptoms.

Women with neurological disorders, current urinary tract infections (UTIs), or a history of recurrent UTIs that could influence pelvic floor function or UI symptoms.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence | 12 weeks
  The International Consultation on Incontinence Questionnaire - Female Lower Urinary Tract Symptoms Long Form (ICIQ-FLUTS-LF) will be used to assess the severity of urinary incontinence.

SECONDARY OUTCOMES:
The Incontinence Quality of Life | 12 Weeks
  The Incontinence Quality of Life questionnaire (I-QOL) will be used to assess the quality of life in patients with urinary incontinence.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Faisalabad, Faisalābad, Punjab Province, Pakistan